CLINICAL TRIAL: NCT07011251
Title: Development of a User Centered Design Approach for Screening, Referral, and Enrollment in Food as Medicine Among Adults
Brief Title: Food Insecurity, Food as Medicine, Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Gustafson (Other)
Responsible Party: Sponsor-Investigator, Alison Gustafson, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 93234; 24FIM1255467 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Food Insecurity; Hypertension
Keywords: Food as medicine
MeSH Terms: conditions — Hypertension | interventions — Food; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The intervention consisted of allocating patients to receive either medically tailored meals or grocery Rx program based on their preferences and resource constraints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Food is Medicine Program Type (Other): Patients were screened for food insecurity either face to face or automated based on standard of care practice at their respective healthcare site. Patients were referred to the study team to utilize a screening decision tool to allocate them to receive either Medically tailored meals or a grocery voucher program. Participants then received their program for 12-weeks. Participants then completed post intervention survey.
  Interventions: Behavioral: Food as Medicine Program; Other: Survey

INTERVENTIONS:
Behavioral: Food as Medicine Program — Grocery Prescription - participants will receive a card loaded with $100 per month to be used on the Instacart Fresh Funds program website/app or a SodaHealth grocery prescription card to be used inside a Kroger or Food City stores. Patients who select grocery delivery where Instacart is not available will receive Food City meals for the same value. or 2) Medically Tailored Meals (MTM) - participants receive approximately 5 frozen meals per week from Mom's Meals that follow an approved diet for those with hypertension. Participants will complete screening questions (screening decision tree attached) after informed consent to determine which food package the participant will receive. The screening decision tree is a tool that asks about kitchen availability for preparing foods, skills, and access to transportation. Depending on how the patient answers they will receive either grocery prescription or MTM for 3-months or 12-weeks.
Other: Survey — Participants answering "no" to assistance but agreeing to the 20-30 minute survey will receive a direct link to a survey related to reasons for not wanting assistance to answer questions at one time point.

SUMMARY:
Development of a user centered design to understand how a tailored food is medicine program based on user preferences and needs improves engagement and clinical outcomes. The study will examine how patients, screened either face to face or through automated for food insecurity, engage in a food is medicine program over 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hypertension in last 12 months
* Experiencing food insecurity as indicated by 2-item Hunger Vital Sign
* English or Spanish speaking
* No plans to move from the area for at least 1 year
* Willing and able to accept text messages
* Free living to the extent that participant has control over dietary intake
* Willing and able to provide written informed consent and participate in all study activities.

Exclusion Criteria:

* Participant in weight research intervention in last 12 months
* Considering bariatric surgery in the next year or prior bariatric surgery
* Lack of safe, stable residence and ability to store meals
* Lack of telephone which can receive text messages
* Pregnancy/breastfeeding or intended pregnancy in the next year
* Known drug or alcohol misuse in the past 2 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Change systolic blood pressure | Baseline and week 12
  captured from the electronic medical record
Change diastolic blood pressure | Baseline and week 12
  captured from the electronic medical record

SECONDARY OUTCOMES:
Change in Dietary Intake | Baseline and week 12
  Dietary intake is captured with the Dietary Screener Questionnaire (DSQ-10). Responses to these dietary intake questions are converted to daily cup equivalent estimates (e.g., 1.2 cups of vegetables per day, 1.1 cups of fruit per day, 2.3 cups of FVs per day) of daily FV intake. The 2020-2025 United States Dietary Guidelines for Americans recommend consuming 2 to 3 cups of vegetables per day and 1.5 to 2 cups of fruit per day.
Change in Nutrition Security | Baseline and week 12
  The one item Gretchen Swanson Nutrition Security question will be asked as follows:In the past month, how often did the participant worry that the food bought wouldn't provide enough nutrients for the family, even if the participant had enough to eat? Response options are never, rarely, sometimes, often, always, don't know
Change in food insecurity | Baseline and week 12
  USDA 6-item food insecurity survey which can be found at this link https://www.ers.usda.gov/topics/food-nutrition-assistance/food-security-in-the-us/survey-tools Scores range from 0-6 with higher scores equating to lower food security

OTHER OUTCOMES:
Number of food insecure participants identified from automated screening | Baseline
Number of participants enrolling in FIM from automated screening | 7 days
Number of food insecure participants identified from face to face screening | Baseline
Number of participants enrolling in FIM from face to face screening | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Alison Gustafson, PhD, MPH, RD, Principal Investigator — University of Kentucky
Locations (1):
- Appalachian Regional Healthcare, Floyd, Kentucky, United States